CLINICAL TRIAL: NCT01612234
Title: Palmitate Metabolism and Insulin Resistance
Brief Title: Saturated Fat Versus Monounsaturated Fat and Insulin Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Craig Lawrence Kien, The Mary Kay Davignon Green and Gold Professor, Depts. of Pediatrics and Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01DK082803 (NIH)
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: humans; lean; obese; saturated fat; monounsaturated fat; insulin sensitivity; inflammation; oxidant stress
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High palmitate or high oleate diet. (Experimental): This is a solid food diet in which vegetable oils are used to create a dietary fat composition similar to the average American/Western diet in which palmitic and oleic acid are ingested in approximately equal amounts (high palmitate diet) or a composition similar to the Mediterranean Diet (low palmitate, high oleate, using hazelnut oil as the source of fat). There are no interventions other than the diet itself.
  Interventions: Dietary Supplement: High palmitate or high oleate diet.
- high palmitate or high oleate diet (Experimental): This is a solid food diet in which vegetable oils are used to create a dietary fat composition similar to the average American/Western diet in which palmitic and oleic acid are ingested in approximately equal amounts (high palmitate diet) or a composition similar to the Mediterranean Diet (low palmitate, high oleate, using hazelnut oil as the source of fat). There are no interventions other than the diet itself.
  Interventions: Dietary Supplement: High palmitate or high oleate diet.

INTERVENTIONS:
Dietary Supplement: High palmitate or high oleate diet. — High palmitate diet composition: Fat, 40.4% kcal; palmitic acid, 16.0% kcal; oleic acid,16.2% kcal. High oleate diet composition: Fat, 40.1% kcal; palmitic acid, 2.4% kcal; oleic acid, 28.8% kcal

SUMMARY:
High intakes of saturated fat are associated with diabetes. Our work has shown that the two most common fatty acids in the North American diet, palmitic acid (saturated fat) and oleic acid (monounsaturated fat) are metabolized differently and have opposite effects on fat burning. The proposed study will examine biochemical and molecular mechanisms for how a high saturated fat diet versus a low saturated fat/high monounsaturated fat diet alters the action of the hormone, insulin, in skeletal muscle.

DETAILED DESCRIPTION:
Palmitic acid (PA), impairs insulin sensitivity in skeletal muscle, and replacing PA in the diet with oleic acid (OA), a monounsaturated fatty acid (FA), may be beneficial. The first objective of this project is to understand the effects on lipid metabolism and skeletal muscle lipid composition, insulin signaling, and inflammatory signaling of two common variations in FA composition of the diet: (1) The typical intake of North America where PA and OA are present in equal proportions (HI PA diet). (2) The Mediterranean FA composition in which PA is much lower and OA much higher (HI OA diet). PA may induce insulin resistance in skeletal muscle cells via its accumulation in lipids within muscle cells and via activation of inflammatory signaling. The second objective of this project is to assess the hypothesis that a high intake of PA will down-regulate its own one-carbon (initial) oxidation, leading to increased inflammatory signaling and decreased insulin signaling. However, there is literature evidence that FA may induce defects in insulin signaling, if FA are not completely oxidized; therefore, the third objective is to assess the hypotheses that a high PA diet may decrease complete oxidation of FA and possibly accelerate initial FA oxidation. A double-masked, cross-over trial of the effects of a high PA diet versus a high OA/low PA diet in 16 overweight or obese subjects and 16 lean subjects (aged 18 - 40 yr) will be conducted to investigate the following Specific Aims:

1. To test the hypothesis that increased intake of PA will cause a decreased rate of [1-13C]-PA oxidation and will be associated with: (a) increased inflammatory signaling, within the muscle and by peripheral blood mononuclear cells; (b) Decreased insulin signaling as characterized by decreased, whole body, peripheral insulin sensitivity (euglycemic/hyperinsulinemic clamp) and, in skeletal muscle, decreased phospho-AKT (Ser473), increased phospho-IRS-1 (Ser636/Ser639), decreased tyrosine phosphorylation of IRS-1, and decreased membrane content of GLUT4.
2. To test the hypothesis that increased intake of PA will cause less complete mitochondrial fatty acid oxidation, perhaps associated with dysfunction of the TCA cycle and increased reactive oxygen species formation. This hypothesis will be tested by measuring whole body and muscle (upper limb) relative rates of oxidation of [13-13C]-PA and [1-13C]-PA and by determining the serum profile of acylcarnitines, the urine concentrations of organic acids, and muscle concentrations of protein carbonyls.
3. To test the hypothesis that a high PA diet will lead to less complete oxidation of FA, less insulin signaling in skeletal muscle in response to a test meal, less whole body insulin sensitivity, increased dysfunction of the TCA cycle, and greater reactive oxygen species formation compared to the results obtained in obese versus lean humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy young adults,
* 18 - 40 years of age

Exclusion Criteria:

* regular aerobic exercise training,
* dyslipidemia, and
* type 2 diabetes or insulin resistance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Whether increased palmitate balance (as measured by intake and the rate of [1-13C]-PA oxidation) causes increased insulin resistance and increased inflammatory signaling by peripheral blood mononuclear cells | up to 4 yr
  Insulin sensitivity, inflammatory signaling, palmitate balance, and incomplete oxidation of palmitate in lean and obese young adults.

SECONDARY OUTCOMES:
We will examine the link between palmitate intake and balance and oxidative stress measured using muscle and peripheral blood markers of oxidative stress and antioxidant responses. | up to 4 yr
  activation of c-Jun N-terminal kinase (JNK) and heme oxygenase 1 in skeletal muscle in response to the diets.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Kien, M.D, Ph.D., Principal Investigator — The University of Vermont
Locations (1):
- The Unversity of Vermont Clinical Research Center at Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Background] Kien CL, Everingham KI, D Stevens R, Fukagawa NK, Muoio DM. Short-term effects of dietary fatty acids on muscle lipid composition and serum acylcarnitine profile in human subjects. Obesity (Silver Spring). 2011 Feb;19(2):305-11. doi: 10.1038/oby.2010.135. Epub 2010 Jun 17. PMID 20559306
- [Background] Kien CL, Bunn JY, Stevens R, Bain J, Ikayeva O, Crain K, Koves TR, Muoio DM. Dietary intake of palmitate and oleate has broad impact on systemic and tissue lipid profiles in humans. Am J Clin Nutr. 2014 Mar;99(3):436-45. doi: 10.3945/ajcn.113.070557. Epub 2014 Jan 15. PMID 24429541
- [Result] Kien CL, Bunn JY, Tompkins CL, Dumas JA, Crain KI, Ebenstein DB, Koves TR, Muoio DM. Substituting dietary monounsaturated fat for saturated fat is associated with increased daily physical activity and resting energy expenditure and with changes in mood. Am J Clin Nutr. 2013 Apr;97(4):689-97. doi: 10.3945/ajcn.112.051730. Epub 2013 Feb 27. PMID 23446891
- [Result] Kien CL, Bunn JY, Poynter ME, Stevens R, Bain J, Ikayeva O, Fukagawa NK, Champagne CM, Crain KI, Koves TR, Muoio DM. A lipidomics analysis of the relationship between dietary fatty acid composition and insulin sensitivity in young adults. Diabetes. 2013 Apr;62(4):1054-63. doi: 10.2337/db12-0363. Epub 2012 Dec 13. PMID 23238293
- [Result] Kien CL, Matthews DE, Poynter ME, Bunn JY, Fukagawa NK, Crain KI, Ebenstein DB, Tarleton EK, Stevens RD, Koves TR, Muoio DM. Increased palmitate intake: higher acylcarnitine concentrations without impaired progression of beta-oxidation. J Lipid Res. 2015 Sep;56(9):1795-807. doi: 10.1194/jlr.M060137. Epub 2015 Jul 8. PMID 26156077
- [Result] Kien CL, Bunn JY, Fukagawa NK, Anathy V, Matthews DE, Crain KI, Ebenstein DB, Tarleton EK, Pratley RE, Poynter ME. Lipidomic evidence that lowering the typical dietary palmitate to oleate ratio in humans decreases the leukocyte production of proinflammatory cytokines and muscle expression of redox-sensitive genes. J Nutr Biochem. 2015 Dec;26(12):1599-606. doi: 10.1016/j.jnutbio.2015.07.014. Epub 2015 Aug 1. PMID 26324406
- See also: Description of Kien Lab at the Division of Endocrinology, Diabetes, and Metabolism, Department of Medicine, The University of Vermont College of Medicine — http://www.uvm.edu/medicine/medicine/endocrinology/?Page=research_lab-kien.html&SM=researchsubmenu.html